CLINICAL TRIAL: NCT04404660
Title: An Open-Label, Multi-Centre, Phase Ib/II Study Evaluating the Safety and Efficacy of AUTO1, a CAR T Cell Treatment Targeting CD19, in Adult Patients With Relapsed or Refractory B Cell Acute Lymphoblastic Leukaemia
Brief Title: A Study of CD19 Targeted CAR T Cell Therapy in Adult Patients With Relapsed or Refractory B Cell Acute Lymphoblastic Leukaemia (ALL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Autolus Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FELIX (AUTO1-AL1); 2019-001937-16 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-05-27 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Relapsed or Refractory B Cell Acute Lymphoblastic Leukemia
Keywords: B cell acute lymphoblastic leukemia; Relapsed B cell acute lymphoblastic leukemia; Refractory B cell acute lymphoblastic leukemia; ALL; AUTO1; CD19-positive CAR T cell
MeSH Terms: conditions — Recurrence; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AUTO1 (Experimental)
  Interventions: Biological: AUTO1

INTERVENTIONS:
Biological: AUTO1 — Following pre-conditioning with chemotherapy (cyclophosphamide and fludarabine) patients will be treated with a total target dose of 410E+6 of CD19-positive CAR T cells as a split dose on Day 1 and on Day 10 (±2 days).
  Other Names: Obecabtagene autoleucel (obe-cel)

SUMMARY:
This is a Phase Ib/II study to evaluate the safety and efficacy of autologous T cells engineered with a chimeric antigen receptor (CAR) targeting CD19 in adult patients with relapsed or refractory B cell acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
This Phase Ib/II, open-label, multi-center, single arm study is designed to evaluate the safety and efficacy of AUTO1 in adult patients with B-cell ALL by determining the overall response rate (ORR).

Adult patients with relapsed or refractory ALL will be enrolled in both phases of the study. Consented patients will go through the following five sequential stages: screening, leukapheresis, pre-conditioning, treatment, and follow-up. All patients will receive a total target dose of 410E+6 of CAR T cells as a split dose on Day 1 and on Day 10 (± 2 days).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older Age 18 years or older
* ECOG performance status of 0 or 1
* Relapsed or refractory B cell ALL
* Patients with Ph+ ALL are eligible if intolerant to TKI, failed two lines of any TKI, or failed one line of second-generation TKI, or if TKI is contraindicated
* Documented CD19 positivity within 1 month of screening
* Phase Ib: Primary Cohort IA: Presence of ≥5% blasts in BM at screening
* Phase Ib: Exploratory Cohort IB: MRD-positive defined as ≥ 1e-4 and <5% blasts in the BM at screening
* Phase II: Primary Cohort IIA: Presence of ≥5% blasts in BM at screening
* Phase II: Cohort IIB: ≥2nd CR or CRi with MRD-positive defined as ≥1e-3 by central ClonoSEQ® NGS testing and <5% blasts in the BM at screening
* Adequate renal, hepatic, pulmonary, and cardiac function

Exclusion Criteria:

* Phase Ib (Cohort IA and Cohort IB) and Phase II (Cohort IIA and Cohort IIB) B-ALL with isolated EM disease
* Diagnosis of Burkitt's leukaemia/lymphoma or CML lymphoid in blast crisis
* History or presence of clinically relevant CNS pathology
* Presence of CNS-3 disease or CNS-2 disease with neurological changes
* Presence of active or uncontrolled fungal, bacterial, viral, or other infection requiring systemic antimicrobials for management
* Active or latent Hepatitis B virus or active Hepatitis C virus
* Human Immunodeficiency Virus (HIV), HTLV-1, HTLV-2, syphilis positive test
* Prior CD19 targeted therapy other than blinatumomab. Patients who have experienced Grade 3 or higher neurotoxicity following blinatumomab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib - Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) occurring after AUTO1 infusion | Up to 24 months
Phase II - Cohort IIA: ORR defined as proportion of patients achieving CR or CRi as assessed by an IRRC. | Up to 24 months

SECONDARY OUTCOMES:
Phase II - Proportion of patients achieving MRD-negative CR by NGS (<1e-4 leukemic cells) | Up to 24 months
Phase II - Complete remission rate | Up to 24 months
Phase II - Response to AUTO1 treatment measured as duration of remission (DOR) | Up to 24 months
Phase II - Response to AUTO1 measured as progression-free survival (PFS). | Up to 24 months
Phase II -Response to AUTO1 treatment measured as overall survival (OS) | Up to 24 months
Phase II - Frequency and severity of AEs and SAEs | Up to 24 months
Phase II - Incidence of severe hypogammaglobulinaemia | Up to 24 months
Phase II - Duration of severe hypogammaglobulinaemia | Up to 24 months
Phase II - Detection of CAR T cells measured by PCR following AUTO1 infusion | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (23):
  - City of Hope National Medical Center, Duarte, California
  - University of California San Diego Health (UCSD), La Jolla, California
  - University of California Davis (UC Davis), Sacramento, California
  - University of California San Francisco (UCSF), San Francisco, California
  - Colorado Blood Cancer Institute (CBCI), Denver, Colorado
  - University of Miami, Miami, Florida
  - H Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - TriStar Centennial Medical Center (SCRI), Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - TTI-Methodist (Texas Transplant Institute) (SCRI), San Antonio, Texas
  - The Medical College of Wisconsin, Milwaukee, Wisconsin
- Spain (3):
  - Fundacio' Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fé, Valencia
- United Kingdom (8):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, Cambridgeshire
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - King's College Hospital, London, Greater London
  - Manchester Royal Infirmary Hospital, Manchester, Greater Manchester
  - Queen Elizabeth University Hospital, Glasgow, Scotland
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - University Hospitals Bristol and Weston NHS Foundation Trust (UHBW), Bristol

REFERENCES:
- [Derived] Jabbour E, Sandhu KS, Shaughnessy P, Logan AC, Abedi M, Shah BD, Bishop MR, Park JH, DeAngelo DJ, Tholouli E, Yallop D, Chaganti S, Hodby K, Barba P, Guerreiro M, Menne T, Shang J, Lao-Sirieix P, Brugger W, Roddie C. Tumor burden-guided dosing contributes to mitigation of immunotoxicities following treatment with obecabtagene autoleucel in adult patients with relapsed/refractory B-cell acute lymphoblastic leukemia. Haematologica. 2026 Jan 8. doi: 10.3324/haematol.2025.288587. Online ahead of print. PMID 41504229
- [Derived] Roddie C, Sandhu KS, Tholouli E, Logan AC, Shaughnessy P, Barba P, Ghobadi A, Guerreiro M, Yallop D, Abedi M, Pantin JM, Yared JA, Beitinjaneh AM, Chaganti S, Hodby K, Menne T, Arellano ML, Malladi R, Shah BD, Mountjoy L, O'Dwyer KM, Peggs KS, Lao-Sirieix P, Zhang Y, Brugger W, Braendle E, Pule M, Bishop MR, DeAngelo DJ, Park JH, Jabbour E. Obecabtagene Autoleucel in Adults with B-Cell Acute Lymphoblastic Leukemia. N Engl J Med. 2024 Dec 12;391(23):2219-2230. doi: 10.1056/NEJMoa2406526. Epub 2024 Nov 27. PMID 39602653